CLINICAL TRIAL: NCT02778126
Title: Disposition of [¹⁴C]LY2606368 Following Intravenous Administration in Patients With Advanced and/or Metastatic Solid Tumours
Brief Title: A Study of Prexasertib (LY2606368) in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15556; I4D-EW-JTJG (Other: Eli Lilly and Company); 2015-003126-13 (EudraCT Number)
Record Dates: First submitted 2016-05-18; First posted 2016-05-19 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — prexasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- [¹⁴C]Prexasertib (Experimental): 170 milligrams (mg) of prexasertib containing approximately 50 μCi [¹⁴C] prexasertib radiotracer administered intravenously (IV) as a 1 hour continuous IV infusion.
  Interventions: Drug: [¹⁴C]Prexasertib
- Prexasertib (Experimental): 105 milligrams per square meter (mg/m²) of prexasertib administered IV as a 1 hour continuous IV infusion once every 14 days (14 day cycles). Treatment may continue until discontinuation criteria are met.
  Treatment for this arm was administered after ¹⁴C administration (¹⁴C was administered during first phase of the study)
  Interventions: Drug: Prexasertib

INTERVENTIONS:
Drug: [¹⁴C]Prexasertib — Administered IV Infusion
  Other Names: [¹⁴C]LY2606368
  Arms: [¹⁴C]Prexasertib
Drug: Prexasertib — Administered IV Infusion
  Other Names: LY2606368
  Arms: Prexasertib

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as Prexasertib (LY2606368) in participants with advanced cancer or cancer that has spread to other parts of the body. This study will involve a single dose of ¹⁴C radiolabelled Prexasertib . This means that a radioactive substance, carbon 14, will be incorporated into the study drug. This will provide information about the study drug and its breakdown products and will help determine how much passes from the blood into urine, feces and expired air. After a minimum 14-day washout period following the [¹⁴C] Prexasertib dose, participants will be allowed to receive continued access to Prexasertib as outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Have a histological or cytological diagnosis of cancer (solid tumour), with clinical or radiologic evidence of locally advanced and/or metastatic disease, for which no life-prolonging therapy exists
* Have the presence of measurable and/or nonmeasurable disease as defined by the Response Evaluation Criteria In Solid Tumours
* Have Body Surface Area (BSA) greater than or equal to (≥)1.62 meter squared (m²) and less than or equal to (≤) 1.90 m²
* Have adequate organ function
* Have a performance status of ≤2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have an estimated life expectancy, in the judgment of the investigator, that will permit the participant to complete 1 full cycle of treatment (beyond the initial [¹⁴C]prexasertib dose)

Exclusion Criteria:

* Have received treatment within 28 days of the initial dose of study drug with an investigational product or non-approved use of a drug or device
* Have serious pre-existing medical conditions (left to the discretion of the investigator)
* Have symptomatic central nervous system (CNS) malignancy or metastasis (screening not required)
* Have current haematologic malignancies or acute or chronic leukaemia
* Have an active fungal, bacterial, and/or known viral infection
* Have participated in a ¹⁴C (carbon) study within the last 6 months prior to screening for this study
* Have a second primary malignancy that in the judgment of the investigator and sponsor may affect the interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09-22; Primary Completion 2017-04-29 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of LY2606368 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Baseline through 120 hours after administration of study drug
Fecal Excretion of LY2606368 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Baseline through 120 hours after administration of study drug
LY2606368 Radioactivity in Expired Air Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Baseline through 120 hours after administration of study drug

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) of LY2606368 and Radioactivity | Predose through 120 hours after administration of study drug
Pharmacokinetics: Area Under the Concentration Time Curve from Time Zero to the Last Measured Concentration (AUC0-tlast) of LY2606368 and Radioactivity | Predose through 120 hours after administration of study drug
Pharmacokinetics: Area Under the Concentration Time Curve from Time Zero to Infinity (AUC0-∞) of LY2606368 and Radioactivity | Predose through 120 hours after administration of study drug
Relative Abundance of LY2606368 As Measured by Percentage of Radioactivity in Feces and Urine | Baseline through 120 hours after administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Liverpool, United Kingdom

REFERENCES:
- See also: Click here for more information about this study: A Study of LY2606368 in Participants With Advanced Cancer — http://www.lillytrialguide.com/en-US/studies/advanced-cancer/JTJG#?postal=